CLINICAL TRIAL: NCT03513757
Title: An Observer-blinded Randomized Study of Propofol Infusion vs Bolus Dexmedetomidine and Propofol Sedation for Pediatric Magnetic Resonance Imaging
Brief Title: Dexmedetomidine and Propofol for Pediatric MRI Sedation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Susan Taylor, Associate Professor, Department of Pediatric Anesthesiology, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CHW 959242-5
Record Dates: First submitted 2018-02-04; First posted 2018-05-02 (Actual); Results first posted 2020-02-21 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Headache; Tumor; Seizure Disorder; Neurofibromatoses; Hydrocephalus; Abdominal Neoplasm; Spine Deformity
MeSH Terms: conditions — Headache; Neoplasms; Epilepsy; Neurofibromatoses; Hydrocephalus; Abdominal Neoplasms | interventions — Propofol; Dexmedetomidine; Glycopyrrolate; Lidocaine; Nitrous Oxide; Sevoflurane

STUDY DESIGN:
Intervention Model Description: observer blinded comparison of propofol with low-dose propofol and dexmedetomidine for pediatric MRI sedation
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The patients and their parents/guardians as well as the blinded observer or investigator who participates in outcomes assessment will be blinded to the drug or drugs administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- propofol (Active Comparator): Each patient will receive 1 mg/kg lidocaine followed by 2 mg/kg propofol IV once prior to continuous propofol infusion for MRI sedation at 200 mcg/kg/min. Dose will be increased by 50 mcg/kg/min up to 300 mcg/kg/min for movement and decreased to 150 mcg/kg/min if no movement after 30 minutes. Additional 1 mg/kg propofol bolus administered at time of each movement. Study to be terminated if movement persists despite above interventions.
  Interventions: Drug: propofol; Drug: Lidocaine 1% Injectable Solution; Drug: Nitrous Oxide; Drug: Sevoflurane
- propofol dexmedetomidine (Experimental): Each patient will receive: 1 mg/kg lidocaine, 2 mg/kg propofol, 4 mcg/kg glycopyrrolate and single dose dexmedetomidine administered prior to scan. Dexmedetomidine dose is dependent on expected duration of scan and will be equal to 1 mcg/kg/hour x duration of scan in hours. 1 mg/kg propofol will be administered for movement up to 2 times. For continued movement after that, begin propofol infusion at 150 mcg/kg/min. Study to be terminated if movement persists despite above interventions.
  Interventions: Drug: propofol; Drug: Dexmedetomidine; Drug: Glycopyrrolate; Drug: Lidocaine 1% Injectable Solution; Drug: Nitrous Oxide; Drug: Sevoflurane

INTERVENTIONS:
Drug: propofol — propofol 2 mg/kg at start of procedure; 2 mg/kg for movement, 150-300 mcg/kg/minute propofol infusion if movement persists
  Other Names: diprivan
Drug: Dexmedetomidine — single dose dexmedetomidine administered at start of sedation in the propofol-dexmedetomidine group. Dosing is based upon anticipated duration of scan from 30 - 75 minutes and will range from 0.5 mic/kg to 1.25 mcg/kg
  Other Names: precedex
  Arms: propofol dexmedetomidine
Drug: Glycopyrrolate — 4 mcg/kg glycopyrrolate will be administered at the start of sedation in the propofol-dexmedetomidine group
  Other Names: Robinul
  Arms: propofol dexmedetomidine
Drug: Lidocaine 1% Injectable Solution — 1 mg/kg intravenous administration prior to propofol administration
  Other Names: Xylocaine 1%
Drug: Nitrous Oxide — Inhalation of nitrous oxide may be used for IV placement
Drug: Sevoflurane — Inhalation of sevoflurane may be used for IV placement
  Other Names: Ultane

SUMMARY:
The purpose of this study is to compare the results of combining two anesthetic medications (dexmedetomidine and propofol) in low doses with a standard dose of a single drug that is commonly used to provide sedation/anesthesia for MRI studies in young children (propofol).

The drugs used for the MRI scan in this study will be chosen randomly. Half the patients will receive small doses of propofol and dexmedetomidine. The other half will receive propofol administered constantly throughout the scan. Other drugs that may be used include sevoflurane and nitrous oxide at the start of the sedation (for placing an intravenous), lidocaine (to reduce the pain of propofol injection) and glycopyrrolate (to prevent the heart rate from decreasing too low. The investigators will record 5 additional blood pressures and heart rates. If additional medications are required to complete the scan, the investigators will administer whatever is necessary. At the end of the study, the investigators will have an observer record the time it takes for participants to spontaneously open eyes , to be able to drink liquids and/or eat and to behave as before the study. Also, it is very important that the investigators find out from participants about changes in behavior, or if eating or sleeping habits were unusual following completion of the study. For that reason, the investigators will call participants in a day or so following the MRI scan.

The investigators expect to recruit 40 children between the ages of 12 and 72 months for the study and hope to have the study completed in December 2018.

DETAILED DESCRIPTION:
The purpose of this study is to compare the results of combining two anesthetic medications (dexmedetomidine and propofol) in low doses with a standard dose of a single drug that is commonly used to provide sedation/anesthesia for MRI studies in young children (propofol).

Recent studies and the FDA have raised concerns that anesthesia for longer than three hours may have effects on behavior and learning. Although investigators do not know if these effects are caused by drugs or the medical condition a child is being treated for, in December 2016, the FDA published the information below regarding anesthesia for children:

General anesthetic and sedation drugs are used to put people into a deep sleep so they do not feel pain during surgery or procedures.

These drugs are usually injected into a vein or breathed in through a mask. General anesthetic and sedation drugs are widely used to ensure the health, safety, and comfort of children and adults undergoing surgery or other procedures.

Recent studies in children suggest that a single, relatively short exposure to general anesthetic and sedation drugs in infants or toddlers is unlikely to have negative effects on behavior or learning. More research is still needed to fully understand how anesthetics might affect brain development, especially longer or repeated exposures and in more vulnerable children. Anesthetic and sedation drugs are necessary for infants, children, and pregnant women who require surgery or other painful and stressful procedures. https://www.fda.gov/Drugs/DrugSafety/ucm532356.htm Research in neonatal and infant animals has demonstrated that sedative and anesthetic agents, like propofol, produce adverse effects on brain development, including loss of brain cells resulting in long-term, possibly permanent changes in learning and behavior. These adverse effects appear to occur mostly after prolonged periods of sedation or anesthesia (generally greater than 3 hours) and when brain development is occurring at a rapid rate (which roughly occurs in children under 3 years of age). It is not known if similar adverse effects occur in humans. Study participants should be advised that the drugs used to accomplish the procedure may have the potential to increase the loss of nerve cells in the developing brain of young child and that the clinical significance of any such changes is not known. There are some animal studies that suggests dexmedetomidine may be better for a growing infant's brain. However, the effects of dexmedetomidine alone or in combination with propofol on the developing brain have not been thoroughly tested to date." The drugs used for the MRI scan in this study will be chosen randomly. Half the patients will receive small doses of propofol and dexmedetomidine. The other half will receive propofol administered constantly throughout the scan. Other drugs that may be used include sevoflurane and nitrous oxide at the start of the sedation (for placing an intravenous), lidocaine (to reduce the pain of propofol injection) and glycopyrrolate (to prevent the heart rate from decreasing too low. Investigators will record 5 additional blood pressures and heart rates. If additional medications are required to complete the scan, investigators will administer whatever is necessary. At the end of the study, an observer will record the time it takes for spontaneous eye opening, to be able to drink liquids and/or eat and to behave as before the study. Also, it is very important that investigators learn in the following day or two how the participant behaved at home; whether eating, behavior and sleeping were unusual. For that reason, the investigator will call the participant a day or so following the MRI scan.

The investigators expect to recruit 70 children between the ages of 12 and 72 months for the study and hope to have the study completed in 2018.

ELIGIBILITY:
Inclusion Criteria:

* All children scheduled for outpatient MRI scans with expected duration of scan between 30 minutes and 75 minutes.

Exclusion Criteria:

* Inpatient status, airway abnormalities, allergy to any study medications, eggs and soy, and mitochondrial disorders.
* All subjects with any cardiac disease or history of cardiac arrhythmias will be excluded.

Ages: 12 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2018-03-04 (Actual); Primary Completion 2018-08-21 (Actual); Study Completion 2018-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan P Taylor, MD, MPH, Principal Investigator — Children's Hospital and Health System Foundation, Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andropoulos DB, Greene MF. Anesthesia and Developing Brains - Implications of the FDA Warning. N Engl J Med. 2017 Mar 9;376(10):905-907. doi: 10.1056/NEJMp1700196. Epub 2017 Feb 8. No abstract available. PMID 28177852
- [Background] Vespasiano M, Finkelstein M, Kurachek S. Propofol sedation: intensivists' experience with 7304 cases in a children's hospital. Pediatrics. 2007 Dec;120(6):e1411-7. doi: 10.1542/peds.2007-0145. PMID 18055659
- [Background] Emrath ET, Stockwell JA, McCracken CE, Simon HK, Kamat PP. Provision of deep procedural sedation by a pediatric sedation team at a freestanding imaging center. Pediatr Radiol. 2014 Aug;44(8):1020-5. doi: 10.1007/s00247-014-2942-z. Epub 2014 May 24. PMID 24859263
- [Background] Mallory MD, Baxter AL, Kost SI; Pediatric Sedation Research Consortium. Propofol vs pentobarbital for sedation of children undergoing magnetic resonance imaging: results from the Pediatric Sedation Research Consortium. Paediatr Anaesth. 2009 Jun;19(6):601-11. doi: 10.1111/j.1460-9592.2009.03023.x. PMID 19645979
- [Background] Mason KP, Zurakowski D, Zgleszewski SE, Robson CD, Carrier M, Hickey PR, Dinardo JA. High dose dexmedetomidine as the sole sedative for pediatric MRI. Paediatr Anaesth. 2008 May;18(5):403-11. doi: 10.1111/j.1460-9592.2008.02468.x. Epub 2008 Mar 18. PMID 18363626
- [Background] Siddappa R, Riggins J, Kariyanna S, Calkins P, Rotta AT. High-dose dexmedetomidine sedation for pediatric MRI. Paediatr Anaesth. 2011 Feb;21(2):153-8. doi: 10.1111/j.1460-9592.2010.03502.x. PMID 21210884
- [Background] Akpinar H, Naziroglu M, Ovey IS, Cig B, Akpinar O. The neuroprotective action of dexmedetomidine on apoptosis, calcium entry and oxidative stress in cerebral ischemia-induced rats: Contribution of TRPM2 and TRPV1 channels. Sci Rep. 2016 Nov 22;6:37196. doi: 10.1038/srep37196. PMID 27872485
- [Background] Boriosi JP, Eickhoff JC, Klein KB, Hollman GA. A retrospective comparison of propofol alone to propofol in combination with dexmedetomidine for pediatric 3T MRI sedation. Paediatr Anaesth. 2017 Jan;27(1):52-59. doi: 10.1111/pan.13041. Epub 2016 Oct 25. PMID 27779360
- [Background] Sikich N, Lerman J. Development and psychometric evaluation of the pediatric anesthesia emergence delirium scale. Anesthesiology. 2004 May;100(5):1138-45. doi: 10.1097/00000542-200405000-00015. PMID 15114210

RESULTS

PARTICIPANT FLOW:
Groups:
- Propofol: Each patient will receive 1 mg/kg lidocaine followed by 2 mg/kg propofol IV once prior to continuous propofol infusion for MRI sedation at 200 mcg/kg/min. Dose will be increased by 50 mcg/kg/min up to 300 mcg/kg/min for movement and decreased to 150 mcg/kg/min if no movement after 30 minutes. Additional 1 mg/kg propofol bolus administered at time of each movement. Study to be terminated if movement persists despite above interventions.
  propofol: propofol 2 mg/kg at start of procedure; 2 mg/kg for movement, 200 mic/kg/minute propofol infusion if movement persists
- Propofol Dexmedetomidine: Each patient will receive: 1 mg/kg lidocaine, 2 mg/kg propofol, 4 mcg/kg glycopyrrolate and single dose dexmedetomidine administered prior to scan. Dexmedetomidine dose is dependent on expected duration of scan and will be equal to 1 mcg/kg/hour x duration of scan in hours. 1 mg/kg propofol will be administered for movement up to 2 times. For continued movement after that, begin propofol infusion at 150 mcg/kg/min. Study to be terminated if movement persists despite above interventions.
  propofol: propofol 2 mg/kg at start of procedure; 2 mg/kg for movement, 200 mic/kg/minute propofol infusion if movement persists
  Dexmedetomidine: single dose dexmedetomidine administered at start of sedation. Dosing is based upon anticipated duration of scan from 30 - 75 minutes and will range from 0.5 mic/kg to 1.25 mic/kg
Period: Overall Study
Arm/Group | Propofol | Propofol Dexmedetomidine
Started | 22 | 18
Completed | 22 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No difference
Groups:
- Propofol: Each patient will receive 1 mg/kg lidocaine followed by 2 mg/kg propofol IV once prior to continuous propofol infusion for MRI sedation at 200 mic/kg/min. Dose will be increased by 50 mic/kg/min up to 300 mic/kg/min for movement and decreased to 150 mic/kg/min if no movement after 30 minutes. Additional 1 mg/kg propofol bolus administered at time of each movement. Study to be terminated if movement persists despite above interventions.
  propofol: propofol 2 mg/kg at start of procedure; 2 mg/kg for movement, 200 mic/kg/minute propofol infusion if movement persists
- Propofol Dexmedetomidine: Each patient will receive: 1 mg/kg lidocaine, 2 mg/kg propofol, 4 mic/kg glycopyrrolate and single dose dexmedetomidine administered prior to scan. Dexmedetomidine dose is dependent on expected duration of scan and will be equal to 1 mic/kg/hour x duration of scan in hours. 1 mg/kg propofol will be administered for movement up to 2 times. For continued movement after that, begin propofol infusion at 150 mic/kg/min. Study to be terminated if movement persists despite above interventions.
  propofol: propofol 2 mg/kg at start of procedure; 2 mg/kg for movement, 200 mic/kg/minute propofol infusion if movement persists
  Dexmedetomidine: single dose dexmedetomidine administered at start of sedation. Dosing is based upon anticipated duration of scan from 30 - 75 minutes and will range from 0.5 mic/kg to 1.25 mic/kg
- Total: Total of all reporting groups
Arm/Group | Propofol | Propofol Dexmedetomidine | Total
Number analyzed (Participants) | 22 | 18 | 40
Age, Continuous [Median (Inter-Quartile Range); unit: months] | 39 [22 to 49] | 26 [22 to 48] | 34 [22 to 47]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 13 | 11 | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 18 | 40

OUTCOME MEASURES:

1. Primary Outcome: Efficiency of Propofol Dexmedetomidine Sedation Compared With Propofol Infusion
Description: Time (minutes) from anesthesia start to readiness for discharge from the department to home or clinic.
Time Frame: through study completion, an average of 2 hours
Measure: Median (Inter-Quartile Range); unit: minutes
Groups:
- Propofol: Each patient will receive 1 mg/kg lidocaine followed by 2 mg/kg propofol IV once prior to continuous propofol infusion for MRI sedation at 200 mcg/kg/min. Dose will be increased by 50 mcg/kg/min up to 300 mic/kg/min for movement and decreased to 150 mcg/kg/min if no movement after 30 minutes. Additional 1 mg/kg propofol bolus administered at time of each movement. Study to be terminated if movement persists despite above interventions.
  propofol: propofol 2 mg/kg at start of procedure; 2 mg/kg for movement, 150-300 mcg/kg/minute propofol infusion if movement persists
Arm/Group | Propofol | Propofol Dexmedetomidine
Number analyzed (Participants) | 22 | 18
minutes | 98 [86 to 115] | 77 [64 to 102]

2. Secondary Outcome: Total Propofol Administered
Description: total propofol administered (mg/kg)
Time Frame: up to 90 minutes
Measure: Median (Inter-Quartile Range); unit: mg/kg
Groups:
- Propofol: Each patient will receive 1 mg/kg lidocaine followed by 2 mg/kg propofol IV once prior to continuous propofol infusion for MRI sedation at 200 mcg/kg/min. Dose will be increased by 50 mcg/kg/min up to 300 mcg/kg/min for movement and decreased to 150 mcg/kg/min if no movement after 30 minutes. Additional 1 mg/kg propofol bolus administered at time of each movement. Study to be terminated if movement persists despite above interventions.
  propofol: propofol 2 mg/kg at start of procedure; 2 mg/kg for movement, 200 mcg/kg/minute propofol infusion if movement persists
Arm/Group | Propofol | Propofol Dexmedetomidine
Number analyzed (Participants) | 22 | 18
mg/kg | 10.6 [9.2 to 12.9] | 3.0 [2 to 3.7]

3. Secondary Outcome: Dexmedetomidine Dose
Description: dexmedetomidine dose (mcg/kg)
Time Frame: up to 90 minutes
Measure: Median (Inter-Quartile Range); unit: mcg/kg
Arm/Group | Propofol | Propofol Dexmedetomidine
Number analyzed (Participants) | 22 | 18
mcg/kg | 0 [0 to 0] | 0.70 [0.70 to 1]

4. Secondary Outcome: Glycopyrrolate Dose
Description: glycopyrrolate dose (mcg/kg)
Time Frame: 5 minutes
Measure: Median (Inter-Quartile Range); unit: mcg/kg
Arm/Group | Propofol | Propofol Dexmedetomidine
Number analyzed (Participants) | 22 | 18
mcg/kg | 0 [0 to 0] | 4.2 [4 to 4.8]

5. Secondary Outcome: Lidocaine Dose
Description: lidocaine dose (mg/kg)
Time Frame: up to 90 minutes
Measure: Median (Inter-Quartile Range); unit: mg/kg
Arm/Group | Propofol | Propofol Dexmedetomidine
Number analyzed (Participants) | 22 | 18
mg/kg | 1.00 [0.97 to 1.03] | 1.00 [0.96 to 1.05]

6. Secondary Outcome: Nitrous Oxide
Description: documentation of use
Time Frame: up to 10 minutes
Measure: Number; unit: participants
Arm/Group | Propofol | Propofol Dexmedetomidine
Number analyzed (Participants) | 22 | 18
participants | 18 | 17

7. Secondary Outcome: Sevoflurane
Description: sevoflurane induction time of 5 minutes
Time Frame: sevoflurane induction time up to 10 minutes
Measure: Number; unit: participants
Arm/Group | Propofol | Propofol Dexmedetomidine
Number analyzed (Participants) | 22 | 18
participants | 18 | 17

8. Secondary Outcome: Eye Opening
Description: minutes from completion of scan to spontaneous eye opening
Time Frame: up to 90 minutes
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Propofol | Propofol Dexmedetomidine
Number analyzed (Participants) | 22 | 18
minutes | 28 [23 to 34] | 3 [2 to 4]

9. Secondary Outcome: Oral/Enteral Intake
Description: minutes from completion of scan to oral/enteral intake
Time Frame: up to 2 hours
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Propofol | Propofol Dexmedetomidine
Number analyzed (Participants) | 22 | 18
minutes | 33 [29 to 42] | 14 [7 to 17]

10. Secondary Outcome: Discharge Ready
Description: minutes from completion of scan to discharge ready
Time Frame: up to 2 hours
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Propofol | Propofol Dexmedetomidine
Number analyzed (Participants) | 22 | 18
minutes | 40 [33 to 53] | 17 [9 to 31]

11. Secondary Outcome: Sleep Pattern
Description: parental observation of deviation from child's normal habit obtained through follow-up phone call
Time Frame: up to 48 hours
Measure: Number; unit: participants
Arm/Group | Propofol | Propofol Dexmedetomidine
Number analyzed (Participants) | 22 | 18
participants | 3 | 2

12. Secondary Outcome: Irritability
Description: behavior deemed inappropriate and a deviation from child's normal though parental observation obtained through follow-up phone call
Time Frame: up to 48 hours
Measure: Number; unit: participants
Groups:
- Propofol Dexmedetomidine: Each patient will receive: 1 mg/kg lidocaine, 2 mg/kg propofol, 4 mcg/kg glycopyrrolate and single dose dexmedetomidine administered prior to scan. Dexmedetomidine dose is dependent on expected duration of scan and will be equal to 1 mcg/kg/hour x duration of scan in hours. 1 mg/kg propofol will be administered for movement up to 2 times. For continued movement after that, begin propofol infusion at 150 mcg/kg/min. Study to be terminated if movement persists despite above interventions.
  propofol: propofol 2 mg/kg at start of procedure; 2 mg/kg for movement, 150-300 mcg/kg/minute propofol infusion if movement persists.
  Dexmedetomidine: single dose dexmedetomidine administered at start of sedation in the propofol-dexmedetomidine group. Dosing is based upon anticipated duration of scan from 30 - 75 minutes and will range from 0.5 mcg/kg to 1.25 mcg/kg.
  Glycopyrrolate: 4 mcg/kg glycopyrrolate will be administered at the start of sedation in the propofol-dexmedetomidine group.
Arm/Group | Propofol | Propofol Dexmedetomidine
Number analyzed (Participants) | 22 | 18
participants | 3 | 0

13. Secondary Outcome: Delirium
Description: Pediatric Anesthesia Emergence Delirium (PAED) score greater than 12 as defined by Sikich and Lerman. 0 = no delirium, 20 = worst possible delirium; 5 categories scored from 0-4 additive for a maximum score of 20. Categories 1-3 are scored the same and categories ar scored inversely as described. 1. Child makes contact with caregiver, 2. child's actions are purposeful, 3. child is aware of his surroundings. For each of these category, score 0 for extremely, 1 for very much, 2 for quite a bit, 3 for just a little, 4 for not at all. The other 2 categories 4. Child is restless and 5 Child is inconsolable are scored as 0 for not at all, 1 for just a little, 2 for quite a bit, 3 for very much, 4 for extremely
Time Frame: up to 24 hours.
Measure: Number; unit: participants
Arm/Group | Propofol | Propofol Dexmedetomidine
Number analyzed (Participants) | 22 | 18
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 48 hours
Arm/Group | Propofol | Propofol Dexmedetomidine
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/18
Other Adverse Events (participants affected / at risk) | 13/22 | 10/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Propofol (N=22) | Propofol Dexmedetomidine (N=18)
respiratory events during induction/anesthesia/recovery (Injury, poisoning and procedural complications) | 10 (10) | 8 (8) — desaturation, cough, breath hold
movement (Injury, poisoning and procedural complications) | 3 (3) | 2 (4) — movement during scan requiring rescan or interruption

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-19): https://cdn.clinicaltrials.gov/large-docs/57/NCT03513757/Prot_SAP_001.pdf